CLINICAL TRIAL: NCT02650635
Title: Phase IB Study Investigating the Tolerability, Immunomodulatory Impacts and, Therapeutic Correlates of the Novel Toll-like Receptor 8 Agonist Motolimod (MOTO) Plus Cyclophosphamide (CTX) Treatment of Advanced Solid Tumors
Brief Title: TLR8 Agonist VTX-2337 and Cyclophosphamide in Treating Patients With Metastatic, Persistent, Recurrent, or Progressive Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: permanently closed per sponsor's request
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1245; NCI-2015-02150 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1245 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2015-12-30; First posted 2016-01-08 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Recurrent Breast Carcinoma; Recurrent Colorectal Carcinoma; Recurrent Melanoma of the Skin; Recurrent Non-Small Cell Lung Carcinoma; Recurrent Pancreatic Carcinoma; Recurrent Renal Cell Carcinoma; Solid Neoplasm; Stage IV Breast Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IV Renal Cell Cancer; Stage IV Skin Melanoma; Stage IVA Colorectal Cancer; Stage IVA Pancreatic Cancer; Stage IVB Colorectal Cancer; Stage IVB Pancreatic Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Carcinoma, Renal Cell | interventions — Cyclophosphamide; pegfilgrastim; VTX-2337

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (CTX, pegfilgrastim, TLR8 agonist VTX-2337) (Experimental): Patients receive cyclophosphamide IV over 30 minutes on day 1, pegfilgrastim SC on day 2, and TLR8 agonist VTX-2337 SC on day -6 of course 1 only and on days 9 and 16. Patients achieving CR, PR, or SD may continue therapy every 21 days for 3 additional courses. Treatment may then continue in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Pegfilgrastim; Other: Pharmacological Study; Drug: TLR8 Agonist VTX-2337

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; HSP-130; Neulasta; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF
Other: Pharmacological Study — Correlative studies
Drug: TLR8 Agonist VTX-2337 — Given SC
  Other Names: Toll-like Receptor 8 Agonist VTX-2337; VTX-2337

SUMMARY:
This phase Ib trial studies the best way of TLR8 Agonist VTX-2337 and cyclophosphamide in treating patients with a solid tumor that has spread from the primary site (place where it started) to other places in the body (metastatic), progressed for a long time (persistent), come back (recurrent), or is growing, spreading, or getting worse (progressed). TLR8 Agonist VTX-2337 may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving TLR8 Agonist VTX-2337 together with cyclophosphamide may be a better treatment for solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the ability of a dosing schedule of cyclophosphamide, pegfilgrastim, and TLR8 agonist VTX-2337 (CyNeuMoto) to reproducibly immunomodulate patients in a manner which enhances the endogenous antitumor effector response.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of this treatment by assessing the adverse events.

II. Best overall response rate, as assessed by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) criteria (irBORR).

III. Duration of tumor response, as assessed by irRECIST (irDOR). IV. Progression-free survival (PFS) as measured by serial imaging studies and assessed by irRECIST.

V. Overall survival, as measured by subject vital status for 36 months following discontinuation of study treatment.

TERTIARY OBJECTIVES:

I. To test the hypothesis that this regimen will prove efficacious as an immunomodulator regardless of the number of prior chemotherapy (chemo) regimens or type of cancer assessed.

II. To evaluate baseline immune status in patients (peripheral blood and intratumoral effector T cells, regulatory T cells, tumoricidal monocytes, and myeloid-derived suppressor cells) as well as the modulatory effects of the treatment upon individual immune components.

III. To correlate treatment-induced immune modulations to clinical outcomes (overall response rate [ORR], progression-free survival [PFS] as determined by immune-related RECIST [irRECIST], and overall survival).

IV. To correlate treatment-induced immune modulations and clinical outcomes to the magnitude of leukopenia (and its surrogate, neutropenia) achieved by the treatment.

OUTLINE:

Patients receive cyclophosphamide intravenously (IV) over 30 minutes on day 1, pegfilgrastim subcutaneously (SC) on day 2, and TLR8 agonist VTX-2337 SC on day -6 of course 1 only and on days 9 and 16. Patients achieving complete response (CR), partial response (PR), or stable disease (SD) may continue therapy every 21 days for 3 additional courses. Treatment may then continue in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic solid tumor, including but not limited to pancreatic adenocarcinoma, breast cancer, melanoma, renal cell carcinoma (RCC), colorectal adenocarcinoma, non-small cell lung cancer, and others approved by the principal investigator
* Persistent, recurrent or progressive disease following at least one prior line of systemic therapy and there is no available therapy likely to improve survival
* Measurable disease with >= 1 target lesion
* White blood cells (WBC) >= 4200/mm^3
* Absolute neutrophil count (ANC) >= 1400/mm^3
* Platelets (PLT) >= 100,000/mm^3
* Lymphocytes >= 700/mm^3
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 1.5 X upper limit of normal (ULN) unless history of Gilbert's syndrome documented prior to first-line treatment of cancer and other liver function tests are within normal limits
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.2 x ULN unless on anticoagulation medication with stable dosing for at least one month; in addition, patient must be able to stop taking medication for up to a week in order to have percutaneous biopsies of tumor tissue performed
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) =< 1.5 x ULN (=< 5 x ULN for patients with liver involvement)
* Creatinine =< ULN or a calculated creatinine clearance of >= 45 ml/min if creatinine is greater than the ULN
* Alkaline phosphatase =< 3 x ULN (=< 5 x ULN if liver or bone involvement)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Willing and able to provide informed written consent
* Willing and able to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study); Note: During the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing and able to return to the consenting institution for follow-up
* Estimated life expectancy >= 84 days (3 months)
* Willing and able to provide samples for correlative research purposes
* If female of child-bearing potential, have a negative pregnancy test =< 14 days prior to registration
* If fertile male or female of child-bearing potential, agree to consistently use a highly effective method of birth control (including birth control pills, barrier device, or intrauterine device) from the time of consent through 4 months following the last dose of study drug

Exclusion Criteria:

* Is pregnant, breastfeeding, or planning a pregnancy
* Known standard therapy for the patient's disease that is potentially curative
* Treatment with any systemic anticancer treatment or an investigational agent within 4 weeks and any radiation within 2 weeks of registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit subject safety or compliance with study requirements
* Active autoimmune disease, defined as any autoimmune condition currently requiring therapy (e.g., systemic lupus erythematosus, multiple sclerosis, inflammatory bowel disease, rheumatoid arthritis)
* History of other invasive malignancy, with the exception of non-melanoma skin cancer and well-excised cervical carcinoma in situ, =< 3 years prior to enrollment unless assessed by the principal investigator as unlikely to compromise subject safety or to interfere with the study's objectives
* Treatment with oral or parenteral corticosteroids dosed greater than 40 mg hydrocortisone daily or its equivalent (e.g., prednisone 10 mg, prednisolone 8 mg, or decadron 3 mg) =< 2 weeks of treatment initiation; or a clinical requirement for ongoing systemic immunosuppressive therapy
* History of central nervous system (CNS) metastases unless previously treated and stable for > 8 weeks prior to study initiation
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive
* Hypersensitivity to pegfilgrastim or Escherichia (E.) coli derived proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Change in pharmacodynamics after TLR8 agonist VTX-2337 alone vs TLR8 agonist VTX-2337+cyclophosphamide | Up to end of course 2 (42 days)
  The pharmacodynamics after TLR8 agonist VTX-2337 alone will be compared to TLR8 agonist VTX-2337+cyclophosphamide to test the hypothesis that TLR8 agonist VTX-2337+cyclophosphamide (course 2) will be significantly more immunomodulatory than TLR8 agonist VTX-2337 alone (course 1 run in dose) in regards to (1) reducing % and absolute numbers of Tregs compared to total lymphocytes; (2) reducing absolute numbers of MDSCs; (3) increasing % of total peripheral T cells activatable to produce IFNg; and (4) increasing % of total peripheral monocytes activatable to produce nitric oxide or express induci

SECONDARY OUTCOMES:
Duration of response, assessed by irDOR, defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the date progression is documented | Up to 36 months
  The distribution of duration of response will be estimated using the method of Kaplan-Meier. Supplemental statistical analysis will include comparison of the duration of response between groups of interest using a Cox proportional hazards model. As an exploratory analysis, will also determine if patients who achieve sustained intratreatment responses (defined as disease stabilization or a maximum objective response unchanged over six cycles of treatment) continue to maintain this response upon cessation of treatment.
Incidence of adverse events of cyclophosphamide and TLR8 agonist VTX-2337, using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 36 months
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns using CTCAE version 4.0.
Overall response rate assessed by irBORR | Up to 36 months
Overall survival (OS) | Time from study entry to death due to any cause, assessed up to 36 months
  The distributions of OS will be estimated using Kaplan-Meier methodology and will be compared between groups of interest using a log-rank test. Supplemental statistical analysis will include comparison of the OS between groups of interest using a Cox proportional hazards model.
PFS as measured by serial imaging studies and assessed by irRECIST | Time from study entry to the first of either progression or death due to any cause, assessed up to 36 months
  The distribution of PFS will be estimated using Kaplan-Meier methodology. Supplemental statistical analysis will include comparison of the PFS between groups of interest using a Cox proportional hazards model.

OTHER OUTCOMES:
Changes in immunomodulation | Baseline to up to day 1 of course 3 (day 63)
  Assessed over time using graphical and statistical methods overall and by treatment course. Changes over time will be assessed using paired t-tests (or the nonparametric equivalent), where changes from baseline and/or course 11 (run-in phase) will be compared to various timepoints of interest post-course 1 (course 2, course 3, etc.). Changes in markers will be assessed by patient groups of interest (i.e. cancer type and the number of prior chemotherapy regimens). Tumor and immune markers will be correlated with clinical endpoints like response, progression-free survival, overall survival, and

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cohen, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States